CLINICAL TRIAL: NCT02114138
Title: Network Analysis of Urinary Molecular Signature Complements Clinical Data to Predict Postoperative Acute Kidney Injury Subtitle: Urinary Molecular and Metabolic Signature of Postoperative Acute Kidney Injury (NavigateAKI)
Brief Title: Network Analysis of Urinary Molecular Signature Complements Clinical Data to Predict Postoperative Acute Kidney Injury
Acronym: NavigateAKI
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400127
Record Dates: First submitted 2014-03-24; First posted 2014-04-15 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury
Keywords: postoperative acute kidney injury; pAKI; stress injury on the kidney; chronic kidney disease; CKD
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical Group: Adults undergoing major in hospital surgery; pathogenesis of perioperative acute kidney injury; urine collection
  Interventions: Procedure: pathogenesis of perioperative acute kidney injury; Diagnostic Test: urine collection
- Healthy Control: Healthy Adult volunteers who are willing to provide a 200 ml urine sample.
  Interventions: Diagnostic Test: urine collection

INTERVENTIONS:
Procedure: pathogenesis of perioperative acute kidney injury — understand pathogenesis of perioperative acute kidney injury in elective and emergent surgery
  Groups: Surgical Group
Diagnostic Test: urine collection — urine collection will be performed on both the control group and hospitalized participants

SUMMARY:
The risk for postoperative acute kidney injury (pAKI), as for any other postoperative complications (PC), comes from a number of interactions between a patient's health before surgery, strength to tolerate surgery and influences on the operating room environment. At this time doctors do not have good tools to predict which patients may be at risk of having this complication. The purpose of this research study is to develop a urine test that can be used to predict the risk for having problems with kidney function after major surgery.

DETAILED DESCRIPTION:
During hospitalization, a urine sample will be collected and additional tests will be added to the daily standard of care blood samples before, during and three times following an elective surgical procedure.

Study participants will complete telephone interviews at 6 and 12 months after discharge from the hospital with a study team member. The telephone interview will consist of a short questionnaire asking about state of health and a health survey.

At the same times of the phone interviews, the study team will mail a urine dipstick that is used to detect any amount of protein in the urine. Study participants will be asked to urinate on dipstick and send it back to the study team in provided shipping material.

Healthy Controls will be enrolled to establish baseline values for kidney health based upon a single urine collection and a brief health questionnaire.

ELIGIBILITY:
Inclusion Criteria for Surgical Group:

* Patients undergoing major in-hospital surgery
* Planned hospital stay of at least 24 hours
* Able to enroll prior to undergoing surgery

Exclusion Criteria for Surgical Group:

* Patients not recruited 4 hours prior to undergoing surgery

Inclusion Criteria for Healthy volunteers:

> 18 years old that elect to serve as a control group

Exclusion Criteria for Healthy volunteers:

Renal Replacement Therapy AKI/CKD Nephrectomy Organ transplant

Any of the following within the last 12 months:

* Stroke/Transient Ischemic Attack
* Heart Attack
* Major Thoracic, abdominal, or Vascular surgery
* Radiation Therapy
* Chemo Therapy
* Immunosuppressive Therapy

IV contrast within the past 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population from which the cohort will be selected among patients undergoing major in-hospital surgery. Healthy Adult Volunteers who meet our enrollment criteria.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2015-07; Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of postoperative acute kidney injury (pAKI) | up to 7 days after surgery.
  PostoperativeAKI is a change outcome of an increase of greater than or equal to 50% of creatinine from initial level prior to surgery until postoperative day 7.

SECONDARY OUTCOMES:
Change from baseline in urine protein biomarkers at 4 hours after surgery | Baseline, 4 hours after surgery
  Change in urine protein biomarkers (urine insulin-like growth factor-binding protein 7 (IGFBP7) and tissue inhibitor of metalloproteinases-2 (TIMP-2)) from prior to surgery (baseline) to four hours after surgery.
Change from baseline in urine protein biomarkers at postoperative day 1 | Baseline, day 1 after surgery
  Change in urine protein biomarkers (urine insulin-like growth factor-binding protein 7 (IGFBP7) and tissue inhibitor of metalloproteinases-2 (TIMP-2)) from prior to surgery (baseline) to postoperative day 1

OTHER OUTCOMES:
All cause mortality | 12 months post-discharge from the hospital.
  Time-to-Event Outcome Measure followed for the duration of study enrollment and specifically measured at 12 months post-discharge from the hospital.
Prolonged mechanical ventilation | Up to 6 months
  Time-to-Event Outcome Measure taken when mechanical ventilation is greater than 48 hours during hospitalization.
chronic kidney disease (CKD) | 12 months post-discharge from the hospital.
  This outcome will be assessed using urinary microalbumin/creatinine ratio (dipstick) mailed to study participants to urinate on and send back to the study team in provided shipping material at 12 months post-discharge from the hospital.
all cause mortality | up to 6 months
  Time-to-Event Outcome Measure followed for the duration of study enrollment and specifically measured at hospital discharge.
all cause mortality | 6 months post-discharge from the hospital.
  Time-to-Event Outcome Measure followed for the duration of study enrollment and specifically measured at 6 months post-discharge from the hospital.
chronic kidney disease (CKD) | 6 months post-discharge from the hospital.
  This outcome will be assessed using urinary microalbumin/creatinine ratio (dipstick) mailed to study participants to urinate on and send back to the study team in provided shipping material at 6 months post-discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Bihorac, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States